CLINICAL TRIAL: NCT00986778
Title: A Comparative Study of Entecavir vs Adefovir Plus Lamivudine vs Combination Entecavir Plus Adefovir in Lamivudine-Resistant Chronic Hepatitis B Chinese Subjects
Brief Title: Entecavir Plus Adefovir in Lamivudine-Resistant Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Objectives Changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-195
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2009-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; entecavir; adefovir; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lamivudine plus Adefovir (Active Comparator)
  Interventions: Drug: Lamivudine; Drug: Adefovir
- Entecavir (Active Comparator)
  Interventions: Drug: Entecavir
- Entecavir plus Adefovir (Experimental)
  Interventions: Drug: Entecavir; Drug: Adefovir

INTERVENTIONS:
Drug: Lamivudine — Tablets, Oral, 100mg, once daily, 48-96 weeks depending on response
  Other Names: Heptotin
  Arms: Lamivudine plus Adefovir
Drug: Entecavir — Tablets, Oral, 1mg, once daily, 48-96 weeks depending on response
  Other Names: Baraclude
  Arms: Entecavir; Entecavir plus Adefovir
Drug: Adefovir — Tablets, Oral, 10mg, once daily, 48-96 weeks depending on response
  Other Names: Hepsera
  Arms: Entecavir plus Adefovir; Lamivudine plus Adefovir

SUMMARY:
Combination therapy with entecavir 1.0 mg plus adefovir 10 mg has superior antiviral activity compared with either entecavir monotherapy 1.0 mg or adefovir 10 mg plus lamivudine 100 mg in Chinese adults with lamivudine-resistant chronic hepatitis B infection

ELIGIBILITY:
Inclusion Criteria:

* CHB HBeAg(+) Subject with Lamivudine treatment history must have LVDr substitution at rtM204V/I
* Naïve to nucleoside/nucleotide analogues except for LVD
* HBV DNA > 17,200 IU/mL
* Compensated liver function
* Serum ALT <10 × ULN

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Evidence of decompensated cirrhosis
* Coinfection with HIV, hepatitis C virus (HCV), or hepatitis D virus (HDV)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with HBV DNA < 50 IU/mL at W48 | Week 48

SECONDARY OUTCOMES:
The proportion of patient with HBV DNA < 50 IU/mL at W 96 | Week 96
Mean reduction of HBV DNA at W 48 & 96 | Week 48 and 96
The proportion of subjects with ALT normalization at W 48 & 96 | Week 48 & Week 96
The proportion of subjects achieved HBeAg loss, seroconversion, HBsAg loss and seroconversion at W48 & 96 | Week 48 & 96
Safety | Week 48 and Week 96
Resistance | Week 48 & Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx